CLINICAL TRIAL: NCT03619564
Title: Chronic Kidney Disease Observational Database - Taiwan
Acronym: CKDOD
Status: Completed | Type: Observational
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: Keto-033-CNI
Record Dates: First submitted 2018-07-24; First posted 2018-08-08 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Chronic Kidney Insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No protein restriction: No protein restriction
- Low protein diet (LPD): LPD: < 0.8 g/kg bodyweight
- Ketoanalogue suppl. very LPD: sVLPD: 0.3-0.4 g/kg bodyweight + keotanalogues

SUMMARY:
The purpose of this study is to determine the effect of a ketoanalogue supplemented very low protein diet on eGFR decline in chronic kidney disease compared to a low protein diet (0.6 g/kg, LPD) or no protein restriction.

DETAILED DESCRIPTION:
An important part of care in chronic kidney disease is an adapted diet. Its most important aspect is protein restriction. The rationale for protein restriction is a reduction of uremic wastes. However, nutritional requirements for protein synthesis limit the maximum extent of protein restriction. To deal with these conflicting targets, a minimum protein intake supplemented with ketoanalogues of amino acids (supplemented very low protein diet, sVLPD) meets the protein needs while reducing uremic waste.

The aim of this explorative, observational study is to determine the effect of sVLPD on eGFR decline compared to a low protein diet (LPD) or no protein restriction.

Data collection The study uses only data from routine health care records. The transfer to the electronic case report form is done by center investigators.

Data entry is monitored monthly for completeness and plausibility. Missing or unusual data will be requested for completion or re-assessment.

In case of high loss to follow up (>10%), low follow up frequency (<90% of patients with <3 visits per year), or greater than 5% missing core data (age, gender, descent, height, weight, history of diabetes and hypertension, blood pressure, serum creatinin, dietary prescription, judgement of compliance), audit visits including source data verification and trainings may be done.

Primary analysis Direct comparison of patients receiving sVLPD or LPD is not meaningful due to the non-interventional design. It is expected that sVLPD patients will have a more advanced stage of CKD, most likely will have higher severity of disease and possibly may have different demographic baseline data. Furthermore, other well-known risk factors for progression of chronic kidney disease like the presence of diabetes mellitus or high blood pressure may affect eGFR decline.

A relevant amount of data is expected to be missing due to the observational nature and the use of data from clinical routine. Furthermore, missing data are unlikely to occur completely at random.

Therefore, missing data will not be imputed but they will be implicitly modeled by a mixed model: mean changes of eGFR from baseline will be analyzed using a restricted maximum-likelihood based repeated measures approach. Analyses will include the fixed, categorical effects of actual treatment, study center, gender, visit time, and baseline variables presence of smoking history, diabetes mellitus, hypertension, and baseline eGFR. Patient will be included as a random factor to the model. Significance tests will use a two-sided α = 0.05.

Secondary analyses Compliance, dietary counselling, use of a nutritional diary, primary diagnosis of CKD, diabetes mellitus, and vegetarian diet will be included to the model described before and analyzed for independent effects or effect modification of the diet.

The approach to the secondary analysis of development of serum urea is similar to the primary analysis.

Cox-regression analysis will be done for time to dialysis initiation or reaching the composite endpoint [>50% eGFR decline or initiation of maintenance dialysis treatment] including the same baseline variables as mentioned for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age >=20 years
* Diagnosis of chronic kidney disease stage 3b to 5 (non-dialysis) according to KDIGO1, i.e. GFR < 45 ml/min/1.73 m².
* Regular dietetic consultancy (at least once a year) for patients with stages 4 and 5 (GFR < 30 ml/min/1.73m²) who are following a LPD or sVLPD.
* Written informed consent according to local regulations

Exclusion Criteria:Hypercalcemia

* Disturbed amino acid metabolism, e.g. phenylketonuria
* A kidney transplant
* Sustained high blood pressure (inadequately controlled (>160 mmHg systolic or >110 mmHg diastolic) despite ≥3 antihypertensive medications)
* Independent life-threatening disease(s), i.e. terminal cancer, AIDS, stage IV heart failure, end stage liver cirrhosis
* Renal insufficiency caused by
* Renal cancer
* Genetic renal diseases, e.g. polycystic kidney disease, congenital nephrotic syndrome
* Hypersensitivity to the active substances or to any of the excipients of the ketoanalogue supplement
* Furthermore, pregnant and breast-feeding patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary nephrologic care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Primary composite endpoint: 50 % eGFR decline or renal replacement therapy [Time Frame: From inclusion to 2 years follow up] | 2 years
  Primary composite endpoint [Time Frame: From inclusion/Patient enrolment to 2 years follow up]. Need for renal replacement therapy or an at least 50% reduction in the estimated glomerular filtration rate (eGFR) compared to time of patient inclusion into the study and after 2 years

SECONDARY OUTCOMES:
Prescribed diet | 2 years
  Prescribed diet (no protein restriction, low protein diet, supplemented very low protein diet), 2 years
Impact of compliance to prescribed protein diet on the eGRF decline | 2 years
  Dietary compliance, 2 years, assessed by consulted dietitian (if available) estimating rated from 0 (not compliant) to 4 (fully compliant); 24 hours urine (if available, urinary urea excretion to assess the actual protein intake in comparison with the prescribed diet [normal diet, LPD, sVLPD)

CONTACTS AND LOCATIONS:
Overall Officials: Hrishikesh Kulkarni, Dr., Study Chair — Fresenius Kabi
Locations (9):
- Taiwan (9):
  - Hualien Tzu Chi Hospital, Hualien City, Hualien County
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Kaohsiung County
  - Keelung Chang Gung Memorial Hospital, Keelung, Keeluing City
  - Taipei Tzu Chi Hospital, Taipei, New Taipei City
  - Shuang Ho Hospital, Taipei, New Taipei City
  - Taichung Veterans General Hospital, Taichung, Taichung City
  - National Cheng Kung University Hospital, Tainan, Tainan County
  - Taipei Veterans General Hospital, Taipei, Taipei City
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No